CLINICAL TRIAL: NCT01592292
Title: A Non-interventional Study for Relative Efficacy Outcome of Rituximab Treatment in RA Patients Who Have Inadequate Response or Have Been Intolerant to a First Anti-TNF Agent
Brief Title: An Observational Study of MabThera (Rituximab) in Patients With Rheumatoid Arthritis And Inadequate Response Or Intolerance to a First Anti-TNF Alpha Therapy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27923
Record Dates: First submitted 2012-04-11; First posted 2012-05-07 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Adalimumab; Etanercept; Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Rituximab: Participants who have inadequate response or were intolerant to the first anti-tumor necrosis factor (anti-TNF) agent in rheumatoid arthritis (RA), receiving rituximab as per physician's discretion for RA treatment were observed for 12 months.
  Interventions: Drug: Rituximab
- Other anti-TNF agent: Participants who have inadequate response or were intolerant to the first anti-TNF agent in RA, receiving other anti-TNF agent, including adalimumab, etanercept and infliximab, as per physician's discretion for RA treatment were observed for 12 months.
  Interventions: Drug: Adalimumab; Drug: Etanercept; Drug: Infliximab

INTERVENTIONS:
Drug: Rituximab — Rituximab as per physician's discretion.
  Other Names: Mabthera
  Groups: Rituximab
Drug: Adalimumab — Adalimumab as per physician's discretion.
  Groups: Other anti-TNF agent
Drug: Etanercept — Etanercept as per physician's discretion.
  Groups: Other anti-TNF agent
Drug: Infliximab — Infliximab as per physician's discretion.
  Groups: Other anti-TNF agent

SUMMARY:
This prospective, multi-center, observational study will evaluate the efficacy and the safety of MabThera (rituximab) in participants with rheumatoid arthritis who have not responded or have been intolerant to a first anti-TNF alpha therapy. Participants have commenced MabThera or an alternative anti-TNF alpha treatment as a second biological therapy. Data will be collected for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/=20 years of age
* Participants with rheumatoid arthritis, who have not responded or have been intolerant to a single anti-TNF alpha therapy and who have initiated MabThera or an alternative anti-TNF alpha therapy

Exclusion Criteria:

* Participants whose first anti-TNF alpha treatment was, or second biological therapy is given as part of a clinical trial studying rheumatoid arthritis
* Participants who have not signed the informed consent form

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with rheumatoid arthritis who have inadequate response or have been intolerant to a first anti-TNF alpha therapy.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- South Korea (10):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Gyeonggi-do
  - Jeju Special Self-Governing Province
  - Jeollabuk-do
  - Seoul
  - Suwon
  - Ulsan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The arm Other anti-TNF agent consisting of participants treated with adalimumab, etanercept and infliximab was divided into individual treatment groups only for the purpose of Participant flow reporting. All other analyses were performed in Rituximab versus Other anti-TNF agent.
Groups:
- Other Anti-TNF Agent: Adalimumab: Participants who have inadequate response or were intolerant to the first anti-TNF agent in RA, receiving adalimumab as per physician's discretion for RA treatment were observed for 12 months.
- Other Anti-TNF Agent: Etanercept: Participants who have inadequate response or were intolerant to the first anti-TNF agent in RA, receiving etanercept as per physician's discretion for RA treatment were observed for 12 months.
- Other Anti-TNF Agent: Infliximab: Participants who have inadequate response or were intolerant to the first anti-TNF agent in RA, receiving infliximab as per physician's discretion for RA treatment were observed for 12 months.
Period: Overall Study
Arm/Group | Rituximab | Other Anti-TNF Agent: Adalimumab | Other Anti-TNF Agent: Etanercept | Other Anti-TNF Agent: Infliximab
Started | 46 | 20 | 13 | 11
Intention to Treat (ITT) Set | 34 (Excluding primary effect evaluation omission.) | 13 | 10 | 8
Standard Population Set (SPS) | 31 (Excluding participants with change of administration drug or suspension of drug administration.) | 10 | 7 | 7
Completed | 40 (Participants who completed 12 months visit.) | 15 | 10 | 10
Not Completed | 6 | 5 | 3 | 1
Not completed — Follow-up loss | 3 | 3 | 1 | 0
Not completed — Withdrew consent | 2 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) set included participants who offered end-point results among the participants who received the study drugs after enrollment and met all inclusion/exclusion criteria.
Groups:
- Other Anti-TNF Agent: Participants who have inadequate response or were intolerant to the first anti-TNF agent in RA, receiving other anti-TNF agent (adalimumab, etanercept or infliximab) as per physician's discretion for RA treatment were observed for 12 months.
- Total: Total of all reporting groups
Arm/Group | Rituximab | Other Anti-TNF Agent | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Customized [Number; unit: participants]
  20-29 years | 0 | 2 | 2
  30-39 years | 4 | 4 | 8
  40-49 years | 7 | 7 | 14
  50-59 years | 6 | 7 | 13
  60-69 years | 15 | 6 | 21
  70-79 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Mean Change From Baseline in DAS28 at Month 6 in Intention to Treat (ITT) Population
Description: DAS28 is calculated from the number of swollen joints and tender joints using the 28-joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and patient's global assessment of disease activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 (minimum score) to 10 (maximum score); higher scores indicated greater affectation due to disease activity. A DAS28 score of less than or equal to (=<) 3.2 = low disease activity, a DAS28 score of >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Month 6
Population: The ITT set included participants who offered end-point results among participants who received study drugs after enrollment and met all inclusion/exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 34 | 31
units on a scale
  Baseline | 6.35 (1.14) | 5.54 (1.14)
  Change at Month 6 | -1.89 (1.73) | -1.80 (1.53)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.3037, ANCOVA — Change in DAS28 at Month 6 was performed using analysis of covariance (ANCOVA) model with baseline DAS28 score and rheumatoid factor (RF) status as covariate values

2. Primary Outcome: Efficacy: Mean Change From Baseline in DAS28 at Month 6 in Standard Population Set (SPS)
Description: as for outcome 1
Time Frame: Baseline and Month 6
Population: The SPS included participants who maintained the secondary biological agent treatment selected for the first time for 6 months among the participants included in the ITT set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 31 | 24
units on a scale
  Baseline | 6.30 (1.18) | 5.47 (1.04)
  Change at Month 6 | -1.74 (1.59) | -1.91 (1.53)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.0951, ANCOVA — Change in DAS28 at Month 6 was performed using ANCOVA model with baseline DAS28 score and rheumatoid factor status as covariate values

3. Secondary Outcome: Efficacy: Mean Change From Baseline in DAS28 at Month 12
Description: as for outcome 1
Time Frame: Baseline and Month 12
Population: Analysis was performed on participants who were administered with secondary biological agent continuously without change or suspension for 12 months. Here, 'n' represents the participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 24 | 17
units on a scale
  Baseline (n=24, 17) | 6.28 (1.27) | 5.49 (0.92)
  Change at Month 12 (n=22, 16) | -2.30 (1.52) | -2.29 (1.36)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.2390, ANCOVA — Change in DAS28 at Month 12 was performed using ANCOVA model with baseline DAS28 score and rheumatoid factor status as covariate values

4. Secondary Outcome: Efficacy: Mean Change From Baseline in Tender Joint Count (TJC) at Month 6 and 12 in Intention to Treat (ITT) Population
Description: TJC is a clinical method to quantify abnormalities in participants with RA. It is associated with the level of pain. The number of tender joints were scored as tender=1 and not tender=0, and counted. A negative change from baseline represents an improvement (a reduction in the number of tender joints).
Time Frame: Baseline, Month 6 and 12
Population: The ITT set included participants who offered end-point results among the participants who received study drugs after enrollment and met all inclusion/exclusion criteria. Here, 'n' represents the participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: number of tender joints
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 34 | 31
number of tender joints
  Baseline (n=34, 31) | 13.38 (7.22) | 8.81 (6.88)
  Change at Month 6 (n=34, 31) | -8.21 (7.54) | -6.32 (7.06)
  Change at Month 12 (n=29, 24) | -9.48 (7.02) | -5.96 (6.40)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.3212, ANCOVA — Change in TJC at Month 6 was performed using ANCOVA model with baseline TJC and baseline rheumatoid factor status as covariate values
Statistical Analysis 2: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.7097, ANCOVA — Change in TJC at Month 12 was performed using ANCOVA model with baseline TJC and baseline rheumatoid factor status as covariate values

5. Secondary Outcome: Efficacy: Mean Change From Baseline in Tender Joint Count (TJC) at Month 6 and 12 in Standard Population Set (SPS)
Description: as for outcome 4
Time Frame: Baseline, Month 6 and 12
Population: The SPS included participants who maintained the secondary biological agent treatment selected for the first time for 6 months among the participants included in the ITT set. Here, 'n' represents the participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: number of tender joints
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 31 | 24
number of tender joints
  Baseline (n=31, 24) | 12.87 (7.32) | 7.79 (5.99)
  Change at Month 6 (n=31, 24) | -7.68 (7.55) | -5.79 (6.17)
  Change at Month 6 (n=26, 20) | -8.62 (6.89) | -5.80 (5.78)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.2444, ANCOVA — Change in TJC at Month 6 was performed using ANCOVA with baseline TJC and baseline rheumatoid factor status as covariate values
Statistical Analysis 2: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.3903, ANCOVA — [p-value comment as in outcome 4, analysis 2]

6. Secondary Outcome: Efficacy: Mean Change From Baseline in Swollen Joint Count (SJC) at Month 6 and 12 in Intention to Treat (ITT) Population
Description: SJC is a clinical method to quantify abnormalities in participants with RA. It reflects the amount of inflamed synovial tissue. The number of swollen joints were scored as swollen=1 and not swollen=0, and counted. A negative change from baseline represents an improvement (a reduction in the number of swollen joints).
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of swollen joints
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 34 | 31
number of swollen joints
  Baseline (n=34, 31) | 11.24 (6.78) | 7.52 (6.63)
  Change at Month 6 (n=34, 31) | -7.00 (6.86) | -5.10 (6.48)
  Change at Month 12 (n-29, 24) | -8.62 (6.52) | -4.29 (5.81)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.5306, ANCOVA — Change in SJC at Month 6 was performed using ANCOVA model with baseline SJC and baseline rheumatoid factor status as covariate values
Statistical Analysis 2: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.2542, ANCOVA — Change in SJC at Month 12 was performed using ANCOVA model with baseline SJC and baseline rheumatoid factor status as covariate values

7. Secondary Outcome: Efficacy: Mean Change From Baseline in Swollen Joint Count (SJC) at Month 6 and 12 in Standard Population Set (SPS)
Description: as for outcome 6
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number of swollen joints
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 31 | 24
number of swollen joints
  Baseline (n=31, 24) | 11.16 (7.10) | 7.13 (6.15)
  Change at Month 6 (n=31, 24) | -6.74 (7.02) | -5.21 (6.35)
  Change at Month 6 (n=26, 20) | -8.31 (6.80) | -5.00 (6.06)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.2549, ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.7644, ANCOVA — [p-value comment as in outcome 6, analysis 2]

8. Secondary Outcome: Efficacy: Mean Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Month 6 and 12 in Intention to Treat (ITT) Population
Description: ESR is an acute phase reactant and a measure of inflammation. A negative change from baseline represents a reduction in inflammation.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimeter/hour (mm/hr)
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 34 | 31
millimeter/hour (mm/hr)
  Baseline (n=34, 31) | 67.00 (27.50) | 60.77 (30.76)
  Change at Month 6 (n=34, 31) | -19.35 (27.03) | -15.55 (33.19)
  Change at Month 12 (n=31, 25) | -20.36 (29.84) | -21.64 (28.16)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.8987, ANCOVA — Change in ESR at Month 6 was performed using ANCOVA model with baseline ESR and rheumatoid factor status as covariate values
Statistical Analysis 2: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.5808, ANCOVA — Change in ESR at Month 12 was performed using ANCOVA model with baseline ESR and rheumatoid factor status as covariate values

9. Secondary Outcome: Efficacy: Mean Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Month 6 and 12 in Standard Population Set (SPS)
Description: as for outcome 8
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 31 | 24
mm/hr
  Baseline (n=31, 24) | 67.55 (28.76) | 61.58 (29.47)
  Change at Month 6 (n=31, 24) | -19.13 (26.96) | -23.21 (31.33)
  Change at Month 12 (n=28, 20) | -21.54 (30.51) | -22.10 (26.11)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.2282, ANCOVA — Change in ESR at Month 6 was performed using ANCOVA model with baseline ESR and baseline rheumatoid factor status as covariate values
Statistical Analysis 2: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.5849, ANCOVA — Change in ESR at Month 12 was performed using ANCOVA model with baseline ESR and baseline rheumatoid factor status as covariate values

10. Secondary Outcome: Efficacy: Mean Change From Baseline in C-reactive Protein (CRP) at Month 6 and 12 in Intention to Treat (ITT) Population
Description: CRP is an inflammation marker. High levels of this protein indicate inflammation in diseases such as RA. A negative change from baseline represents a reduction in inflammation.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 34 | 31
milligram/deciliter (mg/dL)
  Baseline (n=34, 31) | 3.53 (3.07) | 2.56 (2.73)
  Change at Month 6 (n=34, 30) | -1.84 (3.43) | -0.74 (3.25)
  Change at Month 12 (n=31, 25) | -0.69 (6.56) | -1.51 (2.61)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.4900, ANCOVA — Change in CRP at Month 6 was performed using ANCOVA model with baseline CRP and baseline rheumatoid factor status as covariate values
Statistical Analysis 2: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.1826, ANCOVA — Change in CRP at Month 12 was performed using ANCOVA model with baseline CRP and baseline rheumatoid factor status as covariate values

11. Secondary Outcome: Efficacy: Mean Change From Baseline in C-reactive Protein (CRP) at Month 6 and 12 in Standard Population Set (SPS)
Description: as for outcome 10
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 31 | 24
mg/dL
  Baseline (n=31, 24) | 3.53 (3.17) | 2.59 (2.78)
  Change at Month 6 (n=31, 24) | -1.79 (3.56) | -1.63 (2.37)
  Change at Month 12 (n=28, 20) | -0.60 (6.88) | -1.59 (2.73)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.1894, ANCOVA — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.1805, ANCOVA — [p-value comment as in outcome 10, analysis 2]

12. Secondary Outcome: Efficacy: Health Assessment Questionnaire-Disability Index (HAQ-DI) in Intention to Treat (ITT) Population
Description: The HAQ-DI is a participant-completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0 (without any difficulty) to 3 (unable to do). The overall HAQ-DI score is the average of each of the 8 category scores and ranges from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability.
Time Frame: Month 6
Population: The ITT set included participants who offered end-point results among the participants who received study drugs after enrollment and met all inclusion/exclusion criteria. Here number of participants analyzed is the total participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 33 | 30
units on a scale | 0.69 (0.70) | 0.40 (0.48)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.0568, ANCOVA — Change in HAQ-DI at Month 6 was performed using ANCOVA model with baseline rheumatoid factor status as covariate value

13. Secondary Outcome: Efficacy: Health Assessment Questionnaire-Disability Index (HAQ-DI) in Standard Population Set (SPS)
Description: as for outcome 12
Time Frame: Month 6
Population: The SPS included participants who maintained the secondary biological agent treatment selected for the first time for 6 months among the participants included in the ITT set. Here number of participants analyzed is the total participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 30 | 24
units on a scale | 0.73 (0.71) | 0.46 (0.52)
Statistical Analysis 1: Comparison: Rituximab vs Other Anti-TNF Agent; Test type: Superiority or Other; p = 0.1167, ANCOVA — Change in HAQ-DI at Month 6 was performed using ANCOVA model with baseline rheumatoid factor status as covariate value

14. Secondary Outcome: Safety: Number of Participants With Adverse Events (AE), Adverse Drug Reactions (ADR) and Serious Adverse Events
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. ADRs were defined as any response to a drug which was noxious and unintended, and which occurred at dose normally used related to the pharmacological properties. A SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: Baseline up to Month 12
Population: The ITT set included participants who offered end-point results among the participants who received study drugs after enrollment and met all inclusion/exclusion criteria.
Measure: Number; unit: participants
Arm/Group | Rituximab | Other Anti-TNF Agent
Number analyzed (Participants) | 34 | 31
participants
  Adverse events | 8 | 8
  Adverse drug reactions (ADR) | 4 | 5
  Serious adverse events (SAE) | 3 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Description: The ITT set included participants who offered end-point results among the participants who received the study drugs after enrollment and met all inclusion/exclusion criteria.
Arm/Group | Rituximab | Other Anti-TNF Agent
Serious Adverse Events (participants affected / at risk) | 3/34 | 0/31
Other Adverse Events (participants affected / at risk) | 0/34 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=34) | Other Anti-TNF Agent (N=31)
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=34) | Other Anti-TNF Agent (N=31)
Diarrhoea (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.